CLINICAL TRIAL: NCT00461682
Title: A Double-blind, Randomised, Placebo Controlled, Single Dose, Two-period Crossover Study to Investigate the Therapeutic Potential of the TRPV1 Antagonist SB-705498 in Treatment of Subjects With Rectal Hypersensitivity Including Irritable Bowel Syndrome.
Brief Title: Sb-705498 Rectal Pain Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: VRA107438
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Irritable Colon
Keywords: TRPV1 antagonist; Fecal Urgency; rectal pain; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — SB 705498

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-705498

SUMMARY:
SB-705498 has demonstrated efficacy in several preclinical and human experimental pain models. This study will investigate the efficacy of SB-705498 in patients with rectal pain. This will be a double-blind, placebo-controlled, two-way crossover study. 21 patients with faecal urgency (Group 1), and 21 patients with IBS (Group 2) will complete this study.

ELIGIBILITY:
Inclusion Criteria:

* Female/male aged 18-65.
* Women of child bearing potential must use an effective method of contraception
* Faecal urgency as defined by Chan
* ECG, which has no abnormalities
* Normal Clinical labs
* Informed consent and understand protocol requirements
* IBS subjects: Has irritable bowel syndrome (IBS) as defined by Rome II criteria
* Rectal hyperalgesia

Exclusion Criteria:

* Any clinical or biological abnormality found at screen (other than those related to the disease under investigation)
* History of alcohol, substance or drug abuse
* Uncontrolled hypertension
* A history or presence of cardiovascular risk factors
* Participation in a trial within 3 months before the start of the study
* History of allergy
* Unable to withdraw from analgesic medications for their rectal hyperalgesia (opioid-dependent patients can be included if they are willing to withdraw from their opiate medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-01-26; Primary Completion 2007-09-01 (Actual); Study Completion 2007-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 26 January 2007 till 18 September 2007. A total of 21 participants with irritable bowel syndrome (IBS) were planned to be enrolled.
Pre-assignment Details: Due to difficulties with recruitment, only one participant was enrolled in the study; however the participant received only Placebo and not the study drug.
Groups:
- Total Population: Eligible participants were planned to receive oral SB-705498 eight hundred (800) milligrams (mg) once daily or matching Placebo in a randomized manner over two treatment periods once in the study. All participants were planned to be followed-up maximum up to 28 days after the last dose of the study drug.
Period: Overall Study
Arm/Group | Total Population
Started | 1
Completed | 0
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the study drug.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 21 (NA) — Data not reported
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Pain Score to Rectal Distensions at Pre-dose and up to 6 Hours (h) Post-dose of Each Treatment Period
Description: This analysis was performed at 12, 24, 36 and 48 millimeters of mercury (mmHg) which was above the baseline operating pressure threshold. Participants assessed the cough severity and urge to cough using VAS immediately prior to capsaicin challenge. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant. Average of Day -1 and pre-dose was planned as Baseline for VAs assessment. The VAS score was planned to be analyzed on Day-1, Day 1, 2 hours, and 24 hours. Average daily pain scores as captured in participant diary cards were planned to be summarized descriptively and planned to be analyzed. The 11 point pain intensity numerical rating scale ranging from 0 to 10, where 0 represents "No pain" and 10 represents "Worst pain imaginable" was planned to be used for the subjective assessment of the pain.
Time Frame: Baseline (Pre-dose) and up to 6 hours post-dose of each treatment period
Groups:
- Placebo: Eligible participants received matching Placebo during either of the two treatment periods. All participants were planned to be followed-up maximum up to 28 days after the last dose of the Placebo.
- SB-705498: Participants were planned to receive oral SB-705498 800 mg once daily in a randomized manner during either of the two treatment periods. All participants were planned to be followed-up maximum up to 28 days after the last dose of the study drug.
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Visual Analogue Scores for Rectal Distensions for Gas, Urgency to Defecate and Discomfort at Pre-dose and 6 h Post-dose of Each Treatment Period
Description: The VAS scores for assessment of rectal sensation for pain, gas, urgency and discomfort were analyzed separately. Participants assessed the cough severity and urge to cough using VAS immediately prior to capsaicin challenge. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant. Average of Day -1 and pre-dose was planned as Baseline for VAs assessment. The VAS score was planned to be analyzed on Day-1, Day 1, 2 hours, and 24 hours. Average daily pain scores as captured in participant diary cards were planned to be summarized descriptively and planned to be analyzed. The 11 point pain intensity numerical rating scale ranging from 0 to 10, where 0 represents "No pain" and 10 represents "Worst pain imaginable" was planned to be used for the subjective assessment of the pain. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: Baseline (pre-dose) and up to 6 h post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rectal Sensory Thresholds to Thermal Stimulation (Contact Heat Device, Values Reported as in Study) at Pre-dose and 6h Post-dose of Each Treatment Period
Description: Visceral hypersensitivity is defined as reduced pain and discomfort threshold to rectal stimuli. Rectal hypersensitivity was correlated with the degree of rectal hypersensitivity (up-regulation of TRPV-1 receptors) as measured by rectal thermal stimulation. Ongoing rectal pain intensity scale is 11-point numeric rating scale, where 0=Unnoticeable/No Pain, 10=Unbearable/Worst Pain. An average of daily scores over 1 week pre-dose and 1 week post-dose was recorded. Single measurements pre-dose and at hourly intervals within 6 hours post-dose were also recorded. Participants were planned to stay in the hospital for 6h post-dose and were planned to be discharged when physician was satisfied with their medical condition. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant. Participants assessed the cough severity and urge to cough using VAS immediately prior to capsaicin challenge.
Time Frame: Baseline (pre-dose) and 6h post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Peak Pain Intensity Difference (PPID6), as Derived From Maximum Pain Intensity (NRS) Difference From Baseline (Pre-dose on Day 1) by Single Measurement Recorded Over 0-6h of Each Treatment Period
Description: No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant. Change from Baseline (pre-dose) is the value at indicated time-point minus the Baseline value. Average daily pain scores as captured in participant diary cards were planned to be summarized descriptively and planned to be analyzed. The 11 point pain intensity numerical rating scale ranging from 0 to 10, where 0 represents "No pain" and 10 represents "Worst pain imaginable" was planned to be used for the subjective assessment of the pain.
Time Frame: Baseline (pre-dose) and up to 0-6 h of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain Intensity Difference (SPID6), as Derived From Pain Intensity (NRS) Difference From Baseline (Pre-dose on Day 1) by Single Measurement Recorded Over 0-6h Post-dose of Each Treatment Period
Description: Change from Baseline (pre-dose0 is the value at indicated time point minus the Baseline value. Average daily pain scores as captured in participant diary cards were planned to be summarized descriptively and planned to be analyzed. The 11 point pain intensity numerical rating scale ranging from 0 to 10, where 0 represents "No pain" and 10 represents "Worst pain imaginable" was planned to be used for the subjective assessment of the pain. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: Baseline (pre-dose) and up to 0-6 h post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Somatic Heat Pain Thresholds (Hand and Foot) Assessed Pre-dose and 6h Post-dose of Each Treatment Period
Description: Evoked potentials were to be recorded from midline electrodes by placing a ground electrode on temporal lobe region. A low cut off filter with a time constant of 1.06103 and a frequency of 0.15 hertz (Hz) and a high cut off filter of 100Hz was to be applied. The impedance from all electrodes was maintained below 5 ohms (Ω) and the electroencephalogram (EEG) was recorded, digitized at a sampling rate of 500 Hz. Responses from ten stimuli were to be recorded from each participant with the thermode placed over foot and one hand (non-dominant side). The thermode heating rate was set at 70 degree Celsius per second (°C/s) and the cooling rate at 40°C/s. The baseline temperature was 32 °C, destination temperature 51 °C, and stimulus interval approximately of 7 seconds. The participants were allowed to withdraw any time. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: Baseline (pre-dose) and upto 0-6h post-dose for each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Contact Heat-evoked Potentials (CHEPs) - Optional, Assessed Pre-dose and 6h Post-dose of Each Treatment Period
Description: For heat pain threshold measurement, temperature of the thermode was gradually increased from the baseline (32°C) at a rate of 1°C/s. The ramp was stopped and the temperature of the thermode was returned to the Baseline. This was repeated three times. The threshold temperatures and the average value were recorded by the computer. If the thermode temperature reached 50°C without the participant responding, the ramp was stopped and the temperature was returned to baseline automatically to prevent skin injury. This test was performed within two minutes. The respective cut-off temperature is then recorded for that trial. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: Baseline (pre-dose) and 6h post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Defecations Over 24h and Over 1 Week Following a Dose of SB-705498 (Monitored Using Bristol Stool Scoring Diary Kept 1 Week Pre- and 1 Week Post-dose)
Description: Onset associated with change in the frequency and change in the appearance of stools, abnormal stool frequency (>3/day or < 3/week); abnormal stool form (lumpy/hard or loose/watery stool), abnormal stool passage (straining, urgency, or feeling of incomplete evacuation); passage of mucus, and bloating were analyzed over period. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: 7 days pre-dose and 7 days post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Irritable Bowel Syndrome Symptom Severity Score (IBS SSS) Calculated Over Approximately 10 Days Pre- and Post-dose
Description: Participants were rated on a scale based on following parameters - Onset associated with change in the frequency and change in the appearance of stools, abnormal stool frequency (>3/day or < 3/week); abnormal stool form (lumpy/hard or loose/watery stool), abnormal stool passage (straining, urgency, or feeling of incomplete evacuation); passage of mucus, and bloating were analyzed over period. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: 10 days pre-dose and post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Symptom Scoring and Quality of Life Assessments Over Period
Description: Different scales used in this study included HAD, BDI, SF36, Bristol Stool Scoring, IBS QOL and SSS that were used to rate different scores on respective scales. Untreated pain leads to a decrease in daily function capability, social stresses, loss of work, an overall poor quality of life and a burden on healthcare resources. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: Approximately up to 3 months
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Average Daily Pain Scores at Baseline (Pre-dose), 1, 2, 3, 4, 5 and 6h Post-dose for Each Treatment Period
Description: Individual pain scores were collected at screening and pre and post dose during the anorectal physiological assessments. Average daily pain scores as captured in participants' diary cards were summarized descriptively and analyzed. The 11 point pain intensity numerical rating scale ranges from 0 to 10, where 0 represents "No pain" and 10 represents "Worst pain imaginable". This was used for the subjective assessment of the pain over period. No results were reported since the study objectives were not met due to the early study termination and withdrawal of participant.
Time Frame: At Baseline (pre-dose) and each hour post-dose of each treatment period
Arm/Group | Placebo | SB-705498
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately up to 3 months
Description: Safety population included all participants who received at least one dose of the study drug. Due to early termination of the study, only 1 participant was recruited in the study who had one SAE (19 days post placebo) and 0 non-serious AE's is reported.
Groups:
- SB-705498: Participants were planned to receive oral SB-705498 800 milligrams (mg) once daily in a randomized manner during either of the two treatment periods. All participants were planned to be followed-up maximum up to 28 days after the last dose of the study drug.
Arm/Group | Placebo | SB-705498
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | SB-705498 (N=1)
Abdominal (iliac fossa) pain (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.